CLINICAL TRIAL: NCT01757808
Title: A Phase I Study of Ranolazine Acute Administration and Short Term Administration in Pulmonary Arterial Hypertension
Brief Title: A Study of Ranolazine Acute Administration and Short Term Administration in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-0301
Record Dates: First submitted 2012-04-26; First posted 2012-12-31 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; Ranolazine; right ventricle; Safety; cardiopulmonary exercise testing
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Ranolazine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine (Experimental)
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — ranolazine sustained release at a dose of 500mg for one month followed by a dose of 1000mg.
  Other Names: GS-9668
  Arms: Ranolazine
Drug: Placebo — placebo at a dose of 500mg for one month followed by a dose of 1000mg.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety of ranolazine in people with pulmonary arterial hypertension (PAH) and who are receiving 1 or more background PAH therapies: ambrisentan, sildenafil,tadalafil, epoprostenol, treprostinil (IV, SC, inhaled), or iloprost. The primary objective is:

* To estimate the effect of ranolazine administration on acute hemodynamics.
* To assess safety of ranolazine acutely over 6 hrs in the catheterization lab and after 12 weeks of therapy
* To assess changes in right ventricular function after 12 weeks of therapy.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension is a medical disorder in which pressure in the blood vessels going from the right side of the heart to the lungs is higher than normal. The increased blood pressure in the lungs places a strain on the heart. This strain causes the heart to pump less blood into the lungs, causing physical symptoms of shortness of breath and tiredness. The added strain to the heart can cause physical symptoms of swelling in the feet and abdomen. These symptoms can get worse over time due to the decreased pumping ability of the heart.

This study will use a drug called ranolazine. This drug has been approved by the Food and Drug Administration (FDA) to treat chronic angina (chest pain). However, since it has not been approved for use in PAH its use in this study is considered experimental.

ELIGIBILITY:
Inclusion Criteria:

* All subjects age 18-72 yrs will have a diagnosis of PAH. PAH as defined as idiopathic PAH, heritable PAH or PAH associated with collagen vascular disease, congenital heart disease (repaired), or anorexigen use. A history of PAH as defined by hemodynamics at diagnosis by right heart catheterization defined as: mean PAP >25 mmHg with a normal PCWP < 15 mm Hg at rest and a PVR >3 Wood units.
* Baseline 6MW >150 meters
* Patients will be receiving FDA approved PAH monotherapy or dual therapy medications: including, ambrisentan (5,10mg), sildenafil (60-240mg), tadalafil (40mg), epoprostenol, treprostinil, or iloprost at stable doses for >90days.
* Receiving conventional therapy as clinically indicated (oxygen, calcium channel blockers, digoxin) with dose that is unchanged in the preceding 30 days prior to enrollment. This is excluding anticoagulants (warfarin) as the patient's dose may not be stable if the patient is having a cardiac catheterization at baseline within 30 days of enrollment and warfarin is being held.

Exclusion Criteria:

* PAH Category II-IV and Category I associated with all other etiologies: HIV, portopulmonary disease
* All subjects on monotherapy calcium blockers as "calcium blocker responders" irrespective of therapy
* All subjects receiving CY3P4 inducer (i.e. bosentan)
* Subjects with pulmonary hypertension due to significant interstitial lung disease, chronic obstructive pulmonary disease, congestive heart failure, valvular heart disease
* Subjects with (World Health Organization (WHO) functional Class I or Class IV
* Subjects with total lung capacity (TLC) < 60% of predicted
* Subjects with significant obstructive lung disease with FEV1/FVC ratio < 70% of predicted
* Subjects with hypotension defined as systolic arterial pressure < 90 mmHg at baseline
* Subjects with hypertension defined as systolic arterial pressure >140 mmHg at baseline and a diastolic arterial pressure > 90 mmHg despite adequate medical therapy.
* Subjects with impaired renal function as defined as estimated glomerular filtration rate (eGFR) less than 45 mL/min/BSA (where BSA=1.73m2) as calculated by the Modification of Diet in Renal Disease (MDRD) equation:

Patients with eGFR 45-50 mL/min/BSA may be enrolled only after discussion with data safety monitoring board. Patients with eGFR ≥ 50 mL/min/BSA may be enrolled without such a discussion.

* Subjects with liver function tests (transaminases (AST/ALT), total bilirubin, and alkaline phosphatase) >2X normal values
* Subjects with acutely decompensated heart failure requiring hospitalization or medication adjustment or hospitalization for any cause within the previous 30 days prior to screening
* Subjects may not be receiving any other investigational agents
* Subjects with left ventricular ejection fraction <45% or left ventricular shortening fraction <0.2
* Subjects with acute myocardial infarction within 90 days prior to screening
* Subjects taking nitrates for any medical problem
* Subjects with a recent (<180 days) history of pulmonary embolism verified by ventilation/perfusion scan, angiogram or spiral CT scan
* Pregnant or lactating women
* Subjects with a history of current drug abuse including alcohol
* History of gastric bypass surgery
* History of sinus or atrioventricular nodal disease ie. sick sinus syndrome, or second or third degree heart block.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary vascular resistance (PVR) | 12 weeks

SECONDARY OUTCOMES:
Change in CPET (VE/VCO2, PETCO2, peak VO2, peak HR, peak RER, work max (MET or Watt), sub maximum exercise time | 12 weeks
Change in RV echo parameters: 2D, 3D | 12 weeks
Change in 6MWD | 12 weeks
Safety/SAE | 12 weeks
  AE and SAE on study drug and acutely changes in blood pressure and PAP

CONTACTS AND LOCATIONS:
Overall Officials: Mardi Gomberg-Maitland, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Gomberg-Maitland M, Schilz R, Mediratta A, Addetia K, Coslet S, Thomeas V, Gillies H, Oudiz RJ. Phase I safety study of ranolazine in pulmonary arterial hypertension. Pulm Circ. 2015 Dec;5(4):691-700. doi: 10.1086/683813. PMID 26697176